CLINICAL TRIAL: NCT06405035
Title: Dissecting the Role of MIcrobioMe in gastroEsophageal Tumor: a multIdisCiplinary Longitudinal Study
Acronym: MIMETIC
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO-1440
Record Dates: First submitted 2024-03-19; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-03

CONDITIONS: Adenocarcinoma
Keywords: gastroesohageal adenocarcinoma; neoadjuvant chemotherapy; microbiome; radiomics; predictive factor; risk factor; nutrition; genomics; patient-centric model
MeSH Terms: conditions — Adenocarcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples, tissue samples, salivary swabs and fecal samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with resectable gastroesohageal adenocarcinoma: patients with resectable GEA (including Siewert I) which are candidate to receive either peri-op treatments or upfront surgery followed by adjuvant treatments, if recommended.

SUMMARY:
Gastric cancer (GC) is the second leading cause of cancer mortality and remains the fourth common cancer worldwide. Gastric and esophageal cancers treated with curative intent both have a poor prognosis with five-year survival rate varying between 30% and 40% [Hagen]. Therefore, even in the localized or locally advanced (LA) disease, relapse-related death remains a major challenge for curative treatment. Currently, there are several strategies for the curative treatment of GC including perioperative chemotherapy (peri-Op cht), adjuvant chemotherapy and adjuvant chemoradiotherapy. Despite the therapeutic management of localized or LA GC is well established, there is uncertainty about the power of prognostic and predictive factors to tailor anticancer treatments. In addition to that, further investigation is needed to investigate if pre-existing environment factors may act on carcinogenesis and to explore the molecular mechanisms that underlying cancer growth and invasiveness.

DETAILED DESCRIPTION:
Gastric cancer (GC) is the second leading cause of cancer mortality and remains the fourth common cancer worldwide. Gastric and esophageal cancers treated with curative intent both have a poor prognosis with five-year survival rate varying between 30% and 40%. Therefore, even in the localized or locally advanced (LA) disease, relapse-related death remains a major challenge for curative treatment. Currently, there are several strategies for the curative treatment of GC including perioperative chemotherapy (peri-Op cht), adjuvant chemotherapy and adjuvant chemoradiotherapy. Despite the therapeutic management of localized or LA GC is well established, there is uncertainty about the power of prognostic and predictive factors to tailor anticancer treatments. In addition to that, further investigation is needed to investigate if pre-existing environment factors may act on carcinogenesis and to explore the molecular mechanisms that underlying cancer growth and invasiveness.

Gastric carcinogenesis arises as a consequence of a complex interaction between host and environmental factors. It is known that dietary, lifestyle and metabolic factors are implicated in GC. However, although their impact in terms of cancer prevention have been already addressed, we disregard if nutritional disorders and dietary habits may have a potential predictive or prognostic power in LA GC. Therefore, further knowledge is strongly warranted to realize the actual impact of dietary- and lifestyle-factors in GC risk and - conversely - to examine if nutritional disorders are able to negatively impact the outcome of anticancer treatments.

H. pylori infection is the major risk factor associated with non-cardia gastric cancer, and data has emerged with regard to the role of H. pylori eradication for primary prevention of gastric cancer. Smoking has also been implicated as a risk factor for non-cardia cancer. Furthermore, host genetic polymorphisms have an impact on host responses to gastric inflammation and acid secretion, thereby interacting with H. pylori infection and other environmental factors in gastric carcinogenesis. In contrast to non-cardia cancer, H. pylori infection does not play an important role in cardia cancer, with obesity and smoking identified as the main risk factors. Although dietary, lifestyle and metabolic risk factors have been identified, and addressing these lifestyle and metabolic risk factors may contribute to health, the actual impact in modulating cancer response and outcomes is still debated. Results from epidemiological studies reported that dietary factors may play an important role in gastric cancer etiology. Malnutrition is an independent predictor of increased morbidity and mortality. Additionally, weight loss and sarcopenia leads to higher chemotherapy-induced toxicity. In addition, neoadjuvant chemotherapy and chemoradiation therapy, which often worsen a patient's nutritional status, have become a standard treatments. In some cases, anti-cancer treatments may induce weight gain; on the other hand, overweight and obesity represent a risk factor for metabolic syndrome and they may foster disease recurrence. Therefore, it is challenging to estimate how anti-cancer treatments affect nutritional status and vice versa. These serious changes in nutritional status are also associated with marked deterioration in quality of life and can affect the ability to resist infection and recover from surgery. Screening for nutritional risk as early as possible allows for the identification of patients at risk of becoming malnourished. Screening should be done as early as possible, and recent literature suggests that it should be done at diagnosis or at hospital admission; screening should be repeated in the course of treatment for referral for evaluation if needed.Another source of investigation concerns the human microbiome, since microbiota is involved in human health and in several disease. Growing interest in microbiome and immune interaction in oncology lead to the awareness that cancer therapies perturb the microbiota and the host immune response, with resulting dysbiosis. On the other hand, existing evidence supports the hypothesis that gut microbiota can modulate the pharmacological effects and the toxicity profile of anticancer treatments. Therefore, it would be addressed if gut microbiota can shape the efficiency of drugs through several key mechanisms: metabolism, immunomodulation, translocation, enzymatic degradation, reduction of diversity, and ecological variability. Accordingly, microbiome is emerged as a novel target to be explored in different cancer settings. The strongest known risk factor for GC is infection with H.pylori, which drives the development of premalignant lesions (such as gastric atrophy, intestinal metaplasia, and dysplasia) that can lead to gastric cancer. However, although H.pylori is the most common bacterial infection worldwide and colonizes greater than 50% of the global population, only 1%-3% of infected individuals ever develop gastric cancer. In conclusion, although great advances have been made in understanding the complex interplay between the gastric microbiota and H.pylori in the development of gastric inflammation and cancer, further studies are still needed in well-defined human populations to compare differences in the microbiota of H.pylori-infected persons with and without neoplastic lesions. Cross-sectional studies can provide initial insights into microbial associations with cancer; however, reverse effects are a concern, as it is difficult to discern whether carcinogenesis leads to changes in the local microenvironment that creates a new niche for microbes or whether alterations in the microbial population or its functions contribute to carcinogenesis.The study aims to create a unique platform to integrate clinical, biological and imaging data regarding patients with resectable gastric and esophageal adenocarcinoma (GEA). This innovative approach looks at either implementing the data source in resectable GEA and mapping the complex interaction among the aforementioned features (nutrition-microbiome-genomics-radiomics), in order to sharpen the actual precision medicine toward a patient-centric model.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed 8th ed. American Joint Committee on Cancer (AJCC) Stage Ib to Stage III resectable GEA. A multidisciplinary discussion within surgical oncologists, medical oncologists, and radiologist will assess the disease resectability.
2. Signed Written Informed Consent.
3. Patients must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests and all protocol procedures.
4. Males and Females, ages ≥18 years of age.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
6. Have measurable disease based on RECIST 1.1.
7. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion and normal mucosa at baseline and at the time points specified in the Study Procedure Tables.
8. Patients must be medically fit enough to undergo surgery as determined by the treating medical and surgical oncology team.
9. Demonstrate adequate organ function as defined below: Hematologic Absolute neutrophil count (ANC) >/= 1.5 X 10^9/L; Hemoglobin >/= 9.0 g/dL Platelets >/= 100 X 10^9/L prothrombin time (PT)/ international normalized ratio (INR) and partial thromboplastin timePTT </= 1.5 X ULN. Hepatic Total bilirubin </= 1.5 X upper limit normal ULN (isolated bilirubin >1.5 X ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) aspartate aminotransferase AST and alanine aminotransferase ALT Albumin </= 2.5 X ULN 1 >/=2.5 g/dL Renal Creatinine OR Calculated creatinine clearance OR 24-hour urine creatinine clearance </=1.5 X ULN 2 >/= 50 mL/min >/= 50 mL/min.
10. Women are eligible to participate if: non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 mlU/mL and estradiol < 40 pg/mL (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT.
11. The individual methods of contraception and duration should be determined in consultation with the investigator. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of investigational product.
12. Women must not be breastfeeding.
13. Men who are sexually active must use any contraceptive method with a failure rate of less than 1% per year. The investigator shall review contraception methods and the time period that contraception must be followed.
14. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) and azoospermic men do not require contraception.

Exclusion Criteria:

1. Previously or currently receiving cancer therapy (chemotherapy, radiation therapy, immunotherapy, or biologic therapy) or investigational anti-cancer drug.
2. Any major surgery within the last 3 weeks.
3. Stage IV disease at diagnosis.
4. Pregnant or lactating female.
5. Unwillingness or inability to follow the procedures required in the protocol.
6. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
7. Prior malignancy active within the previous 2 years except for patient's prior diagnosis locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast with local control measures (surgery, radiation).
8. Patients with active, known or suspected autoimmune disease. Patients with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
9. Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
10. Patients with a condition requiring systemic treatment with antibiotic or antimycotic medications within 8 weeks from the surgery.
11. Any positive test result for hepatitis B or C virus indicating acute or chronic infection.
12. Known history of testing positive for human immunodeficiency virus or known acquired immunodeficiency syndrome.
13. Patients who are compulsorily detained for treatment of either a psychiatric or physical (infection disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in approximately 130 patients with resectable GEA (from stage IB to III according to TNM VIII edition) who are going to receive upfront surgery or peri-operative management. In the peri-operative cohort, treatments entail a 2 month-period of systemic therapy with FLOT or weakened regimens (i.e. FOLFOX, CAPOX), according to local practice. Surgery will be performed if restaging demonstrates a resectable disease. The choice of access route and type of operation will be chosen according to tumor site and stage, and according to patients' general conditions. Both open and minimally invasive techniques will be used as indicated.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2025-03-08 (Estimated); Study Completion 2026-03-08 (Estimated)

PRIMARY OUTCOMES:
Tumor regression grading (TRG) system | 4 years
  Tumor regression grading (TRG) system, which aims to categorize the amount of regressive changes after cytotoxic treatment mostly refer onto the amount of therapy induced fibrosis in relation to residual tumor or the estimated percentage of residual tumor in relation to the previous tumor site. Commonly used TRGs for upper gastrointestinal carcinomas are the Mandard grading and the Becker grading system. We will apply the Backer grading system.

SECONDARY OUTCOMES:
Pathological complete response (pCR) | 4 years
  Pathological complete response (pCR) is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the resected specimens.
Relapse free survival (RFS) | 4 years
  Relapse free survival (RFS) is defined as the time from random assignment until first recurrence (loco-regional or distant metastasis) or death due to any cause.
Past Nutrition | 4 years
  Past dietary consumption will be measured at baseline using the validated and self-administered food frequency questionnaire (FFQ) developed for the European Prospective Investigation into Cancer and Nutrition Italian section (EPIC) study.
Nutrition risk screening | 4 years
  Nutritional Status will be assessed, using the following Nutrition risk screening - Nutrition Risk Screening 2002 (NRS-2002).
Nutrition status | 4 years
  Nutritional Status will be assessed, using the following Patient Generated Subjective Global Assessment (PG-SGA)
Prognostic Nutrition status | 4 years
  Nutritional Status will be assessed, using the Prognostic nutritional index calculated as follows: 10 x serum albumin (g/dL) + 0.005 x total peripheral lymphocyte count (1000/mcl)
Microbiome | 4 years
  Upper digestive endoscopy with a core biopsy or excisional biopsy will be performed at baseline and one year after surgery .to obtain tissue from tumor tissue and surrounding normal mucosa (1 to 3 cm far from tumor site) for microbiota analysis. The analysis of the microbiota is performed through the use of the most up-to-date bacterial DNA sequencing techniques (Next Generation Sequencing) to guarantee complete and reliable identification of the intestinal microbiota.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Alessandra Cella, MD, Principal Investigator — Istituto Europeo di Oncologia
Locations (1):
- European Institute of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No